CLINICAL TRIAL: NCT02079337
Title: Validation of Subjective Rating Scales Used to Assess Surgical Conditions in Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Matias Vested Madsen, MD, Herlev Hospital
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: NMBVAL2013
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Surgical Conditions; Rating Scales; Laparoscopy; Neuromuscular Blockade; Pneumoperitoneum
MeSH Terms: conditions — Pneumoperitoneum | interventions — Rocuronium; Sugammadex

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Deep NMB (Active Comparator): Videorecordings and subjective ratings of intraabdominal surgical conditions during deep neuromuscular blockade and without neuromuscular blockade
  Interventions: Drug: Rocuronium; Drug: sugammadex; Drug: placebo
- No NMB (Placebo Comparator): Videorecordings and subjective ratings of intraabdominal surgical conditions during no neuromuscular blockade and during deep neuromuscular blockade.
  Interventions: Drug: Rocuronium; Drug: sugammadex; Drug: placebo

INTERVENTIONS:
Drug: Rocuronium
Drug: sugammadex
Drug: placebo

SUMMARY:
Use of neuromuscular blockade (NMB) may improve the surgical work space in patients scheduled for laparoscopic surgical cases (e.g. hysterectomy, ovarian cystectomy, myomectomy). Clinical studies investigating this question often use a numerical or verbal rating scale for subjective evaluation of the surgical workspace. However, no good subjective rating scale have been developed or validated. Neither have possible inter-individual differences in use of such subjective scales been described.

Purpose:

The aim of this study is to validate different subjective rating scales to determine which scale is most useful among surgeons.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years old
* elective gynecologic laparoscopic operation
* can read and understand Danish
* informed consent

Exclusion Criteria:

* BMI > 30 kg/cm2
* known allergy to medications that are included in the project
* severe renal disease, defined by S-creatinine> 0,200 mmol/L, GFR < 30ml/min or hemodialysis)
* neuromuscular disease that may interfere with neuromuscular data
* lactating or pregnant
* impaired liver function
* converting to laparotomy
* perioperative use of neuromuscular blocking agents before randomization
* pneumoperitoneum set to >12 mmHg on the insufflator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Subjective rating scale | Evaluation of video images within a time frame of in average 5 months after surgery
  The subjective rating scale with best possible interobserver agreement described by kappa statistics

SECONDARY OUTCOMES:
Number of correct estimates of level of NMB | Evaluation of video images within a time frame of in average 5 months after surgery
Number of correct estimates of level of NMB according to grade of surgical experience | Evaluation of video images within a time frame of in average 5 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matias V Madsen, MD, Principal Investigator — Herlev Hospital Department of Anethesiology
Locations (1):
- Department of minimal invasive gynecology Aleris-Hamlet Private Hospital, Søborg, Denmark